CLINICAL TRIAL: NCT07263958
Title: HOLLYWOOD: Hemodynamic Evaluation and Management of Pulmonary Hypertension With Inhaled Iloprost in Chronic Obstructive Pulmonary Disease
Brief Title: Hemodynamic Effects of Inhaled Iloprost in PH-COPD (HOLLYWOOD)
Acronym: HOLLYWOOD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Caio Júlio César dos Santos Fernandes, Collaborating Physician, Pulmonary Circulation Group, Heart Institute (InCor), University of São Paulo Medical School, São Paulo, Brazil, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 85760525.5.0000.0068
Record Dates: First submitted 2025-09-05; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Pulmnary Hypertension; COPD; Pulmonary Hypertension Secondary to Lung Disease and/or Hypoxia
Keywords: Pulmonary Hypertension; COPD; Hemodynamics; Prostacyclin Analog; iloprost; Chronic Obstructive Pulmonary Disease (COPD); Group 3 Pulmonary Hypertension; PH-COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Inhaled Iloprost Treatment (Experimental): Participants in this arm will receive inhaled iloprost for a 12-week period. The daily regimen consists of 6 to 9 inhalations, as tolerated. This is a single-group, pre-post study where clinical, exercise, and hemodynamic parameters are assessed at baseline (before treatment) and after 12 weeks to evaluate the efficacy and safety of the intervention.
  Interventions: Drug: Iloprost is a synthetic molecule with pharmacological action

INTERVENTIONS:
Drug: Iloprost is a synthetic molecule with pharmacological action — Ventavis® is the commercial brand name for inhaled iloprost in Brazil.

SUMMARY:
Study Title: A Clinical Study of Inhaled Iloprost for the Treatment of Pulmonary Hypertension in Patients With Chronic Obstructive Pulmonary Disease (HOLLYWOOD)

The goal of this clinical study is to learn if the inhaled drug iloprost is effective and safe for treating pulmonary hypertension (PH) in adult patients who have severe or very severe Chronic Obstructive Pulmonary Disease (COPD).

The main questions it aims to answer are:

Does inhaled iloprost reduce the pressure and resistance in the lung's blood vessels (measured as Pulmonary Vascular Resistance - PVR)?

Does inhaled iloprost improve participants' ability to exercise, measured by how far they can walk in 6 minutes?

What are the side effects and medical problems that participants experience while taking inhaled iloprost?

Researchers will assess changes in participants' health by comparing measurements taken before they start taking inhaled iloprost to measurements taken after 12 weeks of treatment. There is no placebo group in this study.

Participants in this study will:

Use an inhaler to take iloprost 6 to 9 times every day for 12 weeks.

Visit the clinic for checkups at the beginning of the study and after the 12-week treatment period.

Undergo tests including an exercise capacity test (the 6-minute walk test) and heart pressure measurements (hemodynamic tests) before and after the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older.
* Established diagnosis of severe or very severe Chronic Obstructive Pulmonary Disease (COPD), corresponding to GOLD stage 3 or 4.
* Symptomatic Group 3 Pulmonary Hypertension (PH) confirmed by Right Heart Catheterization (RHC) with the following hemodynamic profile at rest:
* Mean Pulmonary Artery Pressure (mPAP) > 35 mmHg.
* Pulmonary Vascular Resistance (PVR) > 5 Wood Units (WU).
* Pulmonary Capillary Wedge Pressure (PCWP) ≤ 15 mmHg.
* Capable of providing written informed consent.

Exclusion criteria:

* History of hypersensitivity to iloprost or other prostacyclin analogs.
* Pregnancy or breastfeeding.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pulmonary Vascular Resistance (PVR) in Wood Units (WU) | Baseline and 12 weeks
  Change in Pulmonary Vascular Resistance (PVR) from baseline to week 12. PVR is a measure of the resistance to blood flow in the pulmonary circulation. It will be measured in Wood Units (WU) and assessed via invasive hemodynamic monitoring (Right Heart Catheterization). A lower PVR indicates improved pulmonary hemodynamics.

SECONDARY OUTCOMES:
Change from Baseline in 6-Minute Walk Distance (6MWD) | Baseline and 12 weeks
  Change in the distance in meteres a participant can walk on a hard, flat surface in 6 minutes. The 6MWD is a measure of exercise capacity.
Change From Baseline in Dyspnea as Measured by the Transitional Dyspnea Index (TDI) Score | Baseline and 12 weeks
  The Transitional Dyspnea Index (TDI) measures changes in dyspnea from a baseline state. The baseline state is established using the Baseline Dyspnea Index (BDI). The TDI score is derived from three categories: functional impairment, magnitude of task, and magnitude of effort. The total score ranges from -9 (major deterioration) to +9 (major improvement). A higher positive score indicates a greater improvement in dyspnea.
Change in Risk of Mortality Stratification | Baseline and 12 weeks
  Change in the patient's risk of mortality as assessed by the COMPERA 2.0 risk assessment model. This model stratifies patients into low, intermediate, or high risk based on a combination of clinical and hemodynamic variables.
Change from Baseline in Mean Right Atrial Pressure (mRAP) | Baseline and 12 weeks
  Change in mean right atrial pressure (mRAP) from baseline to week 12. mRAP reflects right ventricular preload. It will be measured in millimeters of mercury (mmHg) via Right Heart Catheterization.
Change from Baseline in Mean Pulmonary Artery Pressure (mPAP) | Baseline and 12 weeks
  Change in mean pulmonary artery pressure (mPAP) from baseline to week 12. mPAP is a key hemodynamic parameter for monitoring pulmonary hypertension. It will be measured in millimeters of mercury (mmHg) via Right Heart Catheterization.
Change from Baseline in Cardiac Index (CI) | Baseline and 12 weeks
  Change in Cardiac Index (CI) from baseline to week 12. CI is a measure of cardiac performance relative to body size. It will be measured in liters per minute per square meter (L/min/m²) via Right Heart Catheterization. An increase indicates improved cardiac function.
Change from Baseline in Mixed Venous Oxygen Saturation (SvO2) | Baseline and 12 weeks
  Change in mixed venous oxygen saturation (SvO2) from baseline to week 12. SvO2 reflects the balance between systemic oxygen delivery and consumption. It will be measured as a percentage (%) via Right Heart Catheterization.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this article, including clinical, exercise, and hemodynamic data, will be made available to qualified researchers upon reasonable request. A data sharing proposal should be submitted to the corresponding author. The proposal will be reviewed by the study investigators for scientific merit and feasibility. To gain access, data requestors will need to sign a data access agreement and commit to using the data in a manner consistent with the original informed consent provided by the participants.